CLINICAL TRIAL: NCT05084924
Title: Causal Role of Delta-beta Coupling for Goal-directed Behavior in Anhedonia
Brief Title: Investigating the Causal Role of Prefrontal Control in Decision-making in Patients With Anhedonia
Acronym: DEBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-1321; 1K99MH126161-01A1 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder; Anhedonia
Keywords: transcranial Alternating Current Stimulation; Goal-directed behavior; Cross-frequency coupling; Reward-based decision-making
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of three arms of the study: delta-beta tACS, control tACS in theta-gamma, or active sham. Randomization is stratified by SHAPS level such that there are an equal number of participants that are high anhedonia (SHAPS > 33) and low anhedonia (SHAPS <=33).
Who Masked: Participant, Investigator
Masking Description: This study is designed to be double-blind. Participants and the researchers are unaware of each participant's assignment until the completion of all data collection. This is accomplished using randomization codes. Furthermore, this study utilizes an active sham stimulation. This means that the active sham condition includes some stimulation, mimicking the skin sensations associated with tACS. In a previously concluded trial, participants in the delta-beta tACS, theta-gamma tACS, and active sham groups responded similarly to the blinding questionnaire, indicating that the active sham stimulation successfully blinded the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Delta-beta tACS (Experimental): The study is investigating the use of transcranial alternating current stimulation (tACS). The stimulation is delivered at 1 milliampere (mA) zero-to-peak amplitude at the target electrodes and 2 mA zero to-peak amplitude at the return electrode. For the experimental arm, the tACS will be delivered using the cross-frequency stimulation waveform delta-beta (3-20Hz).
  Interventions: Device: Cross-frequency transcranial alternating current stimulation via the NeuroConn Direct Current Stimulator Plus
- Theta-gamma tACS (Active Comparator): This arm serves as an active control where tACS will be delivered using the cross-frequency stimulation waveform theta-gamma (5-50Hz).
  Interventions: Device: Cross-frequency transcranial alternating current stimulation via the NeuroConn Direct Current Stimulator Plus
- Active-sham tACS (Sham Comparator): For active sham stimulation, either delta-beta or theta-gamma stimulation is delivered for 10 seconds and then returns to baseline. This is intended to mimic the skin sensations (e.g., itching, burning, tingling) that are experienced at the onset of stimulation, assisting with blinding the participant's assignment.
  Interventions: Device: Cross-frequency transcranial alternating current stimulation via the NeuroConn Direct Current Stimulator Plus

INTERVENTIONS:
Device: Cross-frequency transcranial alternating current stimulation via the NeuroConn Direct Current Stimulator Plus — Stimulation will be delivered via the NeuroConn Direct Current Stimulator Plus, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research.

SUMMARY:
Investigating whether delta-beta cross-frequency transcranial alternating current stimulation can increase goal-directed behavior in participants with major depressive disorder and elevated symptoms of anhedonia.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to investigate the causal role that delta-beta coupling plays in goal-directed behavior in participants with major depressive disorder (MDD) and symptoms of anhedonia. The participants will perform a reward-based decision-making task. During the task, cross-frequency transcranial alternating current stimulation (tACS) will be delivered at delta-beta frequency, a control-frequency, or an active sham. Electroencephalography will be collected in intermittent resting-state periods. Structural and functional magnetic resonance imaging (MRI) will be collected during the resting-state and during performance of the task.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Have normal to corrected vision
* Willing to comply with all study procedures and be available for the duration of the study
* Speak and understand English
* Low suicide risk as determined by the Columbia Suicide Severity Rating Scale (C-SSRS), and by the Hamilton Depression Rating Scale (HAM-D; less than 3 for the suicidality item).
* Negative pregnancy test for female participants
* Patient Health Questionnaire (PHQ) with 9 items greater than or equal to 10 and a diagnosis of major depressive disorder on the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Attention deficit (hyperactivity) disorder (currently under treatment)
* Neurological disorders and conditions, including, but not limited to: History of epilepsy, seizures (except childhood febrile seizures), dementia, history of stroke, Parkinson's disease, multiple sclerosis, cerebral aneurysm, brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, HIV/AIDS, malignancy, liver or renal impairment)
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* History of current traumatic brain injury
* (For females) Pregnant or breast feeding
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study
* Diagnostic and Statistical Manual of Mental Disorders version 5 diagnosis of present moderate or severe substance use disorder or alcohol use disorder, and past severe substance use disorder or alcohol use disorder, or psychotic disorder within the last 12 months
* Not taking medications for attention deficit (hyperactivity) disorder or benzodiazepines as these medications often produce specific EEG activity that may disrupt our interpretation of the findings
* If major depressive disorder is experienced in episode, the participant must currently be within a depressive episode.
* Contraindications for magnetic resonance imaging (MRI): ferrous metal inside the body, jewelry must be removable, pacemaker or cochlear implant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from 9 to 36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delta-beta tACS | Theta-gamma tACS | Active-sham tACS
Started | 11 | 12 | 12
Completed | 11 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delta-beta tACS | Theta-gamma tACS | Active-sham tACS | Total
Number analyzed (Participants) | 11 | 12 | 12 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 12 | 35
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (12.9) | 27.0 (10.3) | 31.8 (15.6) | 28.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 26
  Male | 2 | 3 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 12 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 9 | 10 | 10 | 29
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in the Percentage of Trials That the Participant Chooses to Perform the Hard Task
Description: In the Expenditure of Effort for Reward Task, participants are faced with a decision on every trial: to choose an easy task with a low effort exertion for a chance at winning a low amount of money or a hard task with a high effort exertion for a chance at winning a greater amount of money. The incentive for the high effort exertion is changed on each trial and the participant gets physically tired from repeated effort exertion. Goal-directed behavior was calculated as the percentage of trials in which the participant decides to perform the high effort exertion. The average of the 4 blocks prior to stimulation served as a baseline (1st hour). The effect of the intervention was the average of the next 8 blocks during stimulation (hours 2 through 3).
Time Frame: Baseline (Hour 1), Stimulation (Hours 2 through 3)
Measure: Mean (Standard Deviation); unit: percentage of trials
Arm/Group | Delta-beta tACS | Theta-gamma tACS | Active-sham tACS
Number analyzed (Participants) | 11 | 12 | 12
percentage of trials | -0.30 (0.15) | -0.22 (0.12) | -0.09 (0.29)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Theta-gamma tACS vs Active-sham tACS; Test type: Superiority; p = 0.049, ANOVA; Main effect of stimulation: F(2,32) = 3.32

2. Secondary Outcome: Change in Coupling Strength Between Low-frequency Prefrontal Signals and High-frequency Posterior Signals
Description: Coupling strength was estimated using the Mean Vector Length calculation between the phase of low-frequency electrical activity in prefrontal electrodes and amplitude of high-frequency activity in posterior cortex. A hybrid signal was created using high-frequency amplitude and low-frequency phase. The magnitude of the average of this signal over time is the coupling strength. Coupling strength was normalized using a z-transformation relative to a null distribution generated by randomly time-shifting the high-frequency data relative to the low-frequency data (z-score). A value of zero represents no coupling. A higher value represents greater coupling strength, which is generally associated with better cognition. Values range from -3 to 3 and a score greater than 1.6 means the coupling is present. The average of the 4 blocks prior to stimulation served as a baseline (1st hour). The effect of the intervention was the average of the next 8 blocks during stimulation (hours 2 through 3).
Time Frame: Baseline (Hour 1), Stimulation (Hours 2 through 3)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Delta-beta tACS | Theta-gamma tACS | Active-sham tACS
Number analyzed (Participants) | 11 | 12 | 12
Z-score | 0.95 (0.68) | -0.97 (1.04) | 0.13 (1.78)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Theta-gamma tACS vs Active-sham tACS; Test type: Superiority; p = 0.004, ANOVA — Main effect of stimulation: F(2,32) = 6.67

ADVERSE EVENTS:
Time Frame: 1 week
Description: Adverse events were systematically assessed after the 3 hour session for all three arms. Each session was approximately 1 week apart. Thus, adverse events were monitored for approximately 1 week.
Arm/Group | Delta-beta tACS | Theta-gamma tACS | Active-sham tACS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/11 | 3/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delta-beta tACS (N=11) | Theta-gamma tACS (N=12) | Active-sham tACS (N=12)
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sleepiness (General disorders) | 0 (0) | 2 (2) | 1 (1)
Trouble Concentrating (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flickering Lights (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Tingling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Burning Sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Local redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Change in mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0)
Ringing in ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05084924/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT05084924/ICF_000.pdf